CLINICAL TRIAL: NCT04626791
Title: A Phase II Study of Modified VR-CAP and Acalabrutinib as First Line Therapy for Transplant-Eligible Patients With Mantle Cell Lymphoma
Brief Title: Modified VR-CAP and Acalabrutinib as First Line Therapy for the Treatment of Transplant-Eligible Patients With Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-LY-1804; NCI-2020-04428 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-LY-1804 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2020-11-03; First posted 2020-11-13 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-08

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — acalabrutinib; Bortezomib; Cyclophosphamide; Cytarabine; Doxorubicin; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Hyaluronoglucosaminidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (modified VR-CAP, acalabrutinib) (Experimental): CYCLES 1, 3, AND 5: Patients receive acalabrutinib PO BID on days 1-21. Patients also receive bortezomib SC on days 1, 8, and 15, rituximab (or rituximab and hyaluronidase human) IV, cyclophosphamide IV, and doxorubicin hydrochloride IV on day 1, and prednisone PO on days 1-5.
  CYCLES 2, 4, AND 6: Patients receive acalabrutinib PO BID on days 1-21. Patients also receive rituximab (or rituximab and hyaluronidase human) IV on day 1 and cytarabine IV on days 1-2.
  Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Acalabrutinib; Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Doxorubicin Hydrochloride; Drug: Prednisone; Biological: Rituximab; Biological: Rituximab and Hyaluronidase Human

INTERVENTIONS:
Drug: Acalabrutinib — Given PO
  Other Names: ACP-196; Bruton Tyrosine Kinase Inhibitor ACP-196
Drug: Bortezomib — Given SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima
Biological: Rituximab and Hyaluronidase Human — Given IV
  Other Names: Rituxan Hycela; Rituximab Plus Hyaluronidase; Rituximab/Hyaluronidase; Rituximab/Hyaluronidase Human

SUMMARY:
This phase II trial investigates how well modified VR-CAP (bortezomib, rituximab, cyclophosphamide, doxorubicin hydrochloride, prednisone, and cytarabine hydrochloride) and acalabrutinib as first line therapy work in treating transplant-eligible patients with mantle cell lymphoma. Modified VR-CAP is a combination of drugs used as standard first line treatment for mantle cell lymphoma. Chemotherapy drugs, such as bortezomib, cyclophosphamide, doxorubicin hydrochloride, and cytarabine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Rituximab is a monoclonal antibody that binds and depletes malignant B cells, by inducing immune responses and direct toxicity. Acalabrutinib blocks a key enzyme which is needed for malignant cell growth in mantle cell lymphoma. Combining modified VR-CAP and acalabrutinib as first line therapy may be more useful against mantle cell lymphoma compared to the usual treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the proportion of complete metabolic responses according to Lugano criteria at the end of study therapy.

SECONDARY OBJECTIVES:

I. To evaluate the safety of this regimen. II. To determine the proportion of subjects proceeding to autologous stem cell transplant (ASCT).

III. To determine the feasibility and results of stem cell mobilization and successful collection.

IV. To determine the progression-free survival (PFS) and overall survival (OS) (event monitoring phase), assessed up to 2 years after registration.

CORRELATIVE RESEARCH OBJECTIVE:

I. To assess minimal residual disease level after 3 and 6 cycles of therapy using the ClonoSEQ (Adaptive Biotechnologies, Seattle, Washington [WA]), and to explore the relationship between radiographic complete response (CR) rate and baseline features.

OUTLINE:

CYCLES 1, 3, AND 5: Patients receive acalabrutinib orally (PO) twice daily (BID) on days 1-21. Patients also receive bortezomib subcutaneously (SC) on days 1, 8, and 15, rituximab (or rituximab and hyaluronidase human) intravenously (IV), cyclophosphamide IV, and doxorubicin hydrochloride IV on day 1, and prednisone PO on days 1-5.

CYCLES 2, 4, AND 6: Patients receive acalabrutinib PO BID on days 1-21. Patients also receive rituximab (or rituximab and hyaluronidase human) IV on day 1 and cytarabine IV on days 1-2.

Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 2 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* No prior therapy for mantle cell lymphoma (MCL)
* MCL in need of systemic therapy, and potentially eligible for ASCT as assessed by the treating physician
* Documented histological confirmation of MCL by local institutional review
* Documented, fludeoxyglucose F-18 (FDG)-avid measurable disease (at least 1 lesion >= 1.5 cm in diameter) as detected by positron emission tomography (PET)/computed tomography (CT) and as defined and includes measurable nodal and extranodal disease sites, or splenomegaly measuring more than 13 cm in vertical length
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, 2
* Absolute neutrophil count (ANC) >= 1000/mm^3 or >= 500/mm^3 if due to lymphomatous marrow or spleen involvement (obtained =< 30 days prior to registration)
* Platelet count >= 100,000/mm^3 or >= 75,000/mm^3 if due to lymphomatous marrow or spleen involvement (obtained =< 30 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (unless documented Gilbert's syndrome, for which total bilirubin =< 3 x upper limit of normal [ULN] is permitted) (obtained =< 30 days prior to registration)
* Aspartate transaminase (AST) =< 3 x ULN (obtained =< 30 days prior to registration)
* Prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) =< 2 x ULN, unless elevated due to a lupus anticoagulant (obtained =< 30 days prior to registration)
* Calculated creatinine clearance must be >= 30 ml/min using the Cockcroft-Gault formula (obtained =< 30 days prior to registration)
* Negative pregnancy test done within =< 14 days prior to registration for women of childbearing potential only
* For women of childbearing potential (WOCBP, defined as premenopausal women capable of becoming pregnant): Must agree to use of highly effective method of birth control during study therapy and until 12 months after last dose of study therapy. NOTE: 'Acceptable' methods are not adequate. Highly effective methods are defined by Clinical Trials Facilitation and Coordination Group [CTFG] as having a failure rate of < 1% per year
* Men must agree to use barrier contraception starting with the first dose of study therapy and through 180 days after completion of study therapy
* Provide informed written consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Hematologic labs must be obtained within =< 14 days of registration
* Willing and able to participate in all required evaluations and procedures in this study protocol
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information

Exclusion Criteria:

* Prior systemic treatment for mantle cell lymphoma. Short course of steroids (=< 7 days) for symptom management or localized radiation is permissible, as long as measurable disease outside of the radiation field exists
* Peripheral neuropathy or neuropathic pain of grade 2 or worse as assessed by the investigator
* Prior exposure to bortezomib or a BTK inhibitor
* Prior anthracycline exposure unless cumulative prior exposure is under 150 mg per square meter
* Requiring anticoagulation with warfarin or equivalent vitamin k antagonist
* Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenia purpura)
* Active bleeding or history of bleeding diathesis (e.g. hemophilia or von Willebrand disease)
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer
* Requiring treatment with a proton pump inhibitor. Examples include: dexlansoprazole, esomeprazole, lansoprazole, omeprazole, pantoprazole, rabeprazole, or therapeutic class equivalents

  * Note: H2-receptor agonists are not exclusionary
* History of allergic reactions attributed to acalabrutinib, cytarabine, bortezomib, boron, or any of the other agents administered as part of the therapeutic regimen in this study
* Active systemic fungal, bacterial, viral, or other infection that is worsening (defined as increasing signs/symptoms of infection during screening) or, requires intravenous antibiotic therapy
* Active or chronic uncontrolled hepatitis B or hepatitis C infection. Patients with positive hepatitis B core antibody positive require negative polymerase chain reaction (PCR) prior to enrollment. Hepatitis B surface antigen positive or PCR positive patients will be excluded. Patients with hepatitis C must have negative hepatitis C virus (HCV) ribonucleic acid (RNA) for inclusion
* Co-morbid systemic illnesses or other severe concurrent disease (including major surgery within 2 weeks) which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Known to be human immunodeficiency virus (HIV) positive since antiretroviral therapy has a potential for drug interactions with acalabrutinib
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure or low cardiac ejection fraction (New York Heart Association [NYHA] class 3-4 or ejection fraction [EF] < 45%), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 2 years prior to registration. EXCEPTIONS: Non-melanotic skin cancer localized prostate cancer, or carcinoma-in-situ of the breast or cervix. NOTE: If there is a history or prior malignancy, patients must not be receiving other specific treatment for their cancer
* Pregnant and/or breastfeeding
* Has difficulty with or is unable to swallow oral medication, or has significant gastrointestinal disease that would limit absorption of oral medication
* Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening. unless directly due to MCL Involvement by endoscopic or histologic evaluation
* Major surgical procedure within 28 days of first dose of study drug. NOTE: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug
* Concurrent participation in another therapeutic clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-08-03 (Actual); Primary Completion 2024-08-03 (Estimated); Study Completion 2028-08-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of complete responses to therapy (complete metabolic response [CMR]) | At completion of study treatment
  Measured according to Lugano criteria. A success is defined as a CMR as the objective status at the end of treatment. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. 9% confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Minimal residual disease (MRD) rate | Up to completion of study treatment
  Measured by flow. MRD results will be reported descriptively, and explored for correlation with clinical factors and patient outcomes.
MRD rate | Up to completion of study treatment
  Measured by sequencing. MRD results will be reported descriptively, and explored for correlation with clinical factors and patient outcomes.
Incidence of adverse events | Up to 30 days post-treatment
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be reported.
Progression-free survival | From the date of registration to the date of progression (or relapse),or death due to any cause, whichever comes first, assessed at 2 years post-registration
  The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Overall survival | From registration to death due to any cause, assessed at 2 years post-registration
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Feasibility of stem cell collection | Up to completion of study treatment
  The proportion of patients successfully collecting at least 2 x 10^6 CD34 cells/kg pt body weight will be calculated and reported.
Successful proceeding to autologous stem cell transplant (ASCT) | Up to completion of study treatment
  The proportion of patients successfully proceeding to ASCT will be calculated and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Smith, Principal Investigator — Academic and Community Cancer Research United
Locations (7):
- United States (7):
  - Ochsner NCI Community Oncology Research Program, New Orleans, Louisiana
  - Metropolitan-Mount Sinai Medical Center, Minneapolis, Minnesota
  - Mount Sinai Hospital, New York, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin